CLINICAL TRIAL: NCT04736121
Title: A Prospective, Multicenter, Open-label Single Arm Study Evaluating the Safety & Efficacy of Selective Internal Radiation Therapy Using SIR-Spheres® Y-90 Resin Microspheres on DoR & ORR in Unresectable Hepatocellular Carcinoma Patients
Brief Title: Selective Internal Radiation Therapy (SIRT) Using SIR-Spheres® Y-90 Resin Microspheres on DoR & ORR in Unresectable Hepatocellular Carcinoma Patients
Acronym: DOORwaY90
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sirtex Medical (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STX2001
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Unresectable Hepatocellular Carcinoma; BCLC Stage A Hepatocellular Carcinoma; BCLC Stage B Hepatocellular Carcinoma; BCLC Stage C Hepatocellular Carcinoma
Keywords: Unresectable hepatocellular carcinoma; HCC; Unresectable metastatic liver tumor; SIR-Spheres microspheres; Y-90 resin microspheres; Barcelona Clinic Liver Cancer; BCLC; SIRT (Selective Internal Radiation Therapy); Liver cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: A pivotal, prospective, multicenter, open-label single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Open-label Single Arm (Experimental): Open-label single arm study evaluating treatment with hepatic arterial injection of SIR-Spheres.
  Interventions: Device: Resin microspheres containing yttrium-90 (Y-90)

INTERVENTIONS:
Device: Resin microspheres containing yttrium-90 (Y-90) — Biocompatible resin microspheres are an injectable permanent implant and preferentially placed into the distal microvascular supply of tumors to provide direct irradiation of tissue and destruction of the microvascular bed. Spheres contain yttrium-90 (Y-90) and are a size between 20 and 60 microns in diameter.

SUMMARY:
The objective of this pivotal study is to evaluate the safety and effectiveness of SIRT using SIR-Spheres Y-90 resin microspheres as first-line treatment for local control of HCC in patients with Barcelona Clinic Liver Cancer (BCLC) stage A, B1, B2, and C.

SIR-Spheres consist of biocompatible resin microspheres containing yttrium-90 (Y-90), with a size between 20 and 60 microns in diameter. Y-90 is a high-energy pure beta-emitting isotope with no primary gamma emission.

SIR-Spheres are indicated for the local tumor control of unresectable hepatocellular carcinoma (HCC) in patients with Barcelona Clinic Liver Cancer (BCLC) stage A, B1 and B2, maximal single lesion size of 8 cm, no macrovascular invasion, well-compensated liver function and good performance status. It is also indicated for the treatment of unresectable metastatic liver tumors from primary colorectal cancer with adjuvant intra-hepatic artery chemotherapy (IHAC) of Floxuridine (FUDR).

DETAILED DESCRIPTION:
The investigation is a pivotal, prospective, multicenter, open-label single arm study evaluating treatment with hepatic arterial injection of SIR-Spheres.

Up to 100 subjects will be treated (up to 150 consented) at up to 30 clinical sites in the United States.

The population for this study includes patients diagnosed with HCC BCLC stage A, B1, B2, and C with maximal single lesion size of ≤ 8cm and who are not considered suitable for treatment by resection or eligible for ablation at time of study entry.

ELIGIBILITY:
Inclusion Criteria:

1. Willing, able, and mentally competent to provide written informed consent
2. Age 18 or older at the time of consent
3. All tumors must be measurable by CT or MRI according to localized mRECIST
4. Life expectancy ≥ 6 months (to allow for adequate completion of study procedures and collection of data)
5. Diagnosis of HCC with Liver Imaging Reporting and Data System (LIRADS) 4 or 5 or by histology
6. Treatment-naïve patients or patients who have developed a new lesion following one of these prior locoregional treatments:

   1. Liver resection with negative pathologic margins, no microvascular invasion, and no recurrence at resection margins for at least 6 months post-treatment and no new lesions within 6 months of liver resection
   2. Ablation of a single ≤3cm lesion with no recurrence of the treated lesion for at least 6 months post-treatment
7. BCLC stage A, B1, B2, and C with maximal single tumor size of ≤8 cm and sum of the maximal tumor dimensions of ≤12 cm with the entire tumor burden expected to be treatable within the perfused volume
8. At least one lesion ≥1 cm in diameter (long axis) measured according to mRECIST criteria by CT or MRI
9. Child-Pugh score of A5 or A6 at baseline
10. Eastern Cooperative Oncology Group (ECOG) performance score of ≤1 at baseline
11. Adequate blood count, liver enzymes, and renal function at baseline

    1. Platelet count >50,000/microliter (patients may not receive a platelet transfusion or growth factors to increase the platelet count so that the patient may be eligible for the study)
    2. White Blood Cell (WBC) ≥ 3 x 10^9/L
    3. Hemoglobin > 8.5 g/dL
    4. Aspartate transaminase (AST) & Alanine transaminase (ALT) < 5 x upper limit normal
    5. Bilirubin ≤ 2.0 mg/dL
    6. Albumin > 3.0 g/dL
    7. International normalized ratio (INR) ≤ 2.0
    8. Glomerular filtration rate (GFR) > 50
12. Negative serum pregnancy test at baseline
13. Life expectancy of > 3 months without any active treatment

Exclusion Criteria:

1. Patients eligible for ablation or resection for their malignancy, in the opinion of the investigator, at the time of screening
2. Prior systemic anti-cancer therapy (including immunotherapy and/or targeted therapy), radiotherapy or use of other investigational agents for the treatment of HCC
3. Intrahepatic arteriovenous shunting (arteriovenous shunting resulting from a biopsy is allowed but must be embolized during the pre-treatment mapping procedure)
4. Incompetent biliary duct system, prior biliary intervention or a compromised Ampulla of Vater
5. Planned localized cancer treatment to the liver, other than the study treatment, throughout the duration of the study.
6. Planned systemic cancer treatment throughout the duration of the study
7. Patients with portal vein thrombosis
8. Patients with extrahepatic disease
9. Patients with contraindications to angiography and selective visceral catheterization
10. Evidence of extrahepatic collateral supply to the tumor
11. Evidence of potential delivery of mean radiation dose > 30 Gy to the lungs (single treatment)
12. Evidence of any detectable 99m Tc-macroaggregated albumin (99m Tc-MAA) flow outside of the liver in the abdomen, after application of established angiographic techniques to stop or mitigate such flow (e.g., placing catheter distal to gastric vessels or coiling)
13. Evidence that < 33% of the total liver volume is disease-free and will be spared SIR-Spheres treatment
14. Prior liver resection and/or liver transplant, with exception for patients with prior resection who meet inclusion criterion 6a
15. Female patients who are pregnant, breastfeeding, or premenopausal and unwilling to use an effective method of contraception through the 1-year follow-up; males unwilling to use effective method of contraception for 30 days post-procedure
16. Medical history of clotting disorders
17. Underlying pulmonary disease requiring chronic oxygen therapy
18. Evidence of portal hypertension with ascites as seen on cross-sectional imaging or any history of prior variceal bleeding within 6 months prior to screening
19. Concurrently enrolled in another study unless it is an observational, noninterventional study
20. Active infection (hepatitis B (HBV) infection with ongoing HBV treatment and successfully treated hepatitis C infection are allowed)
21. History of other cancer with current active treatment
22. Patients with drug or alcohol dependency (within 6 months prior to study entry) in the opinion of the investigator
23. History of severe allergy or intolerance to contrast agents, narcotics, or sedatives
24. Any condition that, in the opinion of the investigator, would interfere with safe delivery of the study treatment or with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 9 months
  ORR uses a localized version of modified Response Evaluation Criteria in Solid Tumors ("localized mRECIST") criteria and best response through 9 months, in patients treated with SIR-Spheres Y-90 resin microspheres.
Duration of Response (DoR) | 12 months
  The interval from first time of response (complete response (CR) or partial response (PR)) until disease progression (PD) as defined by localized mRECIST criteria.

SECONDARY OUTCOMES:
Grade ≥ 3 toxicity (CTCAE v5.0) | 2 months and 6 months
  The severity of the adverse event should be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Incidence of liver resection | Post-procedure follow-up: 1, 2, 4, 6, 9, 12, 24 months
  Liver resection as noted on follow-up case report form.
Incidence of liver transplant | Post-procedure follow-up: 1, 2, 4, 6, 9, 12, 24 months
  Liver transplant as noted on follow-up case report form.
Quality of life metrics - FACT-Hep Questionnaire | Pre-procedure, 2, 4, 6, 9, and 12 months
  Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) questionnaire
Quality of life metrics - EQ-5D-5L Questionnaire | Pre-procedure, 2, 4, 6, 9, and 12 months
  EuroQol 5 Dimension 5 Level (EQ-5D-5L) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Armeen Mahvash, M.D., Principal Investigator — M.D. Anderson Cancer Center; S. Cheenu Kappadath, Ph.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (22):
- United States (22):
  - University of California Los Angeles - Ronald Reagan Medical Center, Los Angeles, California
  - Providence St. Joseph Hospital, Orange, California
  - University of California Irvine, Orange, California
  - Miami Cardiac and Vascular Institute at Baptist Hospital, Miami, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Columbia University CUIMC/NYPH, New York, New York
  - University of North Carolina - Chapel Hill Medical Center, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center CTO, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Clinical Research Institute and Methodist Hospital, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Inland Imaging, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahvash A, Chartier S, Turco M, Habib P, Griffith S, Brown S, Kappadath SC. A prospective, multicenter, open-label, single-arm clinical trial design to evaluate the safety and efficacy of 90Y resin microspheres for the treatment of unresectable HCC: the DOORwaY90 (Duration Of Objective Response with arterial Ytrrium-90) study. BMC Gastroenterol. 2022 Mar 28;22(1):151. doi: 10.1186/s12876-022-02204-1. PMID 35346070